CLINICAL TRIAL: NCT02093507
Title: Effectiveness of Parent's Manipulation in Newborn With Metatarsus Adducts.a Randomized Controlled Trial
Brief Title: Effectiveness of Parent's Manipulation in Newborn With Metatarsus Adducts. a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SI 172/2
Record Dates: First submitted 2014-03-16; First posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Foot Deformity Congenital
Keywords: newborn; foot deformity congenital
MeSH Terms: conditions — Foot Deformities, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- parents manipulation (Experimental): parents manipulation
  Interventions: Other: parents manipulation
- no manipulation (No Intervention): no manipulation

INTERVENTIONS:
Other: parents manipulation — parents perform manipulation the child foot to correct the deformity
  Arms: parents manipulation

SUMMARY:
The purpose of this study is to determine whether the result of parent's feet manipulation compared with nonmanipulated group within first 6 months of life and observe spectrum of the disease within this period.

DETAILED DESCRIPTION:
The newborn with metatarsus adducts are included in the study and divide in 2 groups by random.Group A with parents'manipulation of the foot and group B without manipulation of the foot.The parents'foot manipulation is trained by pediatric orthopedic surgeons to correct the deformity.The effectiveness of the manipulation is measured by percentage of no deformity of the foot in newborn after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* newborn with Metatarsus adducts.

Exclusion Criteria:

* 1. criteria were included newborns with associated life threatening conditions. 2. congenital or musculoskeletal problems.(ie;arthrogryposis multiplex congenita,skeletal dysplasia) 3. mental retardation. 4. cognitive impairment. 5. parents incooperative. 6. difficult to follow up patients.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
evidence of no foot deformity of newborn | 6 month
  in the group of parents manipulation or in the group without parents manipulation ,for the period of 6 months the outcomes measurement will be done to assess the evidence of foot deformity remaining by pediatric orthopedic surgeons, the outcomes will be the percentage of success or success rate

SECONDARY OUTCOMES:
the statistical significant difference between sex and duration from disease to cure | 6 month
  the sex and duration of treatment are the secondary outcomes measurement to evaluate the statistical difference between both groups

OTHER OUTCOMES:
the satisfaction score | 6 month
  the satisfaction score of parents to manipulate their children feet

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr.Kamolporn - Kaewpornsawan, M.D., Principal Investigator — Department of orthopaedic surgery,faculty of medicine Siriraj Hospital,Mahidol University,Banfkok,Thailand
Locations (1):
- Siriraj hospoital, Bangkoknoi, Bangkok, Thailand